CLINICAL TRIAL: NCT01943591
Title: DELTA Trial: Does Embolization With Larger Coils Lead to Better Treatment of Aneurysms Trial
Acronym: DELTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: DePuy Synthes (Industry); Johnson & Johnson Medical Companies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE13.092
Record Dates: First submitted 2013-09-12; First posted 2013-09-17 (Estimated); Results first posted 2020-01-22 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2018-12

CONDITIONS: Cerebral Aneurysm
Keywords: treatment trial; cerebral aneurysm; randomized; coils; endovascular; Aneurysm; Intracranial Aneurysm; Vascular Diseases; Cardiovascular Diseases; Intracranial Arterial Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm; Vascular Diseases; Cardiovascular Diseases; Intracranial Arterial Diseases; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 15-caliber platinum coils (Experimental): Endovascular embolization coiling using 15-caliber platinum coils
  Interventions: Device: Endovascular coiling with standard 10-caliber platinum coils or 15-caliber platinum coils
- 10-caliber coils (Active Comparator): Endovascular embolization coiling using standard 10-caliber platinum coils
  Interventions: Device: Endovascular coiling with standard 10-caliber platinum coils or 15-caliber platinum coils

INTERVENTIONS:
Device: Endovascular coiling with standard 10-caliber platinum coils or 15-caliber platinum coils — Embolization using 15-caliber platinum coils or standard 10-caliber platinum coils.

SUMMARY:
Endovascular treatment with platinum coils is safe and effective in preventing rebleeding of intracranial aneurysms. Unfortunately, endovascular treatment of aneurysms with coils has been associated with incomplete occlusion at initial treatment (remnant) or at follow-up (recurrence). This in some studies has been as high as 20%. While many such aneurysm remnants or recurrences exhibit benign behavior, many require retreatment to prevent future hemorrhage.

A recent randomized controlled trial of aneurysm coiling revealed that aneurysms between 2 and 9.9 mm diameter were more likely to have an improved angiographic and composite clinical outcome when treated with hydrogel-coated coils, an improvement inferred to result from higher packing density afforded by hydrogel expansion(1). The use of hydrogel coils is associated with technical difficulties related to expansion and limited time for deployment. The investigators theorize that similar results could be achieved by using more voluminous bare platinum coils, leading to improved packing density compared to smaller caliber coils, and thus result in lower incidence of remnants or residuals. The relationship between packing densities and composite clinical endpoints having never been shown in a robust fashion, the investigators therefore propose a randomized clinical trial opposing coiling with soft 15-caliber coils to 10-caliber bare platinum coils in aneurysms varying in size from 3 to 9.9 mm.

To test the hypothesis that 15-caliber coiling systems are superior to standard 10-caliber coils in achieving better composite outcomes, the investigators propose the DELTA trial: Does Embolization with Larger coils lead to better Treatment of Aneurysms trial, a randomized controlled blinded trial with 2 subgroups of 282 patients each, 564 total:

Subgroup 1: Coiled with a maximum proportion of 15-caliber coils as conditions allow Subgroup 2: Coiled with 10-caliber coils.

ELIGIBILITY:
Inclusion Criteria:

* At least one ruptured or unruptured aneurysms with a dimension ≥ 10 mm (longest axis)
* for ruptured lesions, patients should be in World Federation of Neurosurgical Societies (WFNS) grade < IV.
* The anatomy of the lesion is such that endovascular treatment is possible with both types of coils (not necessarily certain or probable)
* Patient is 18 or older
* Life expectancy is more than 2 years (able to complete follow-up)

Exclusion Criteria:

* Patients with planned treatment of an associated cerebral arteriovenous malformations
* When parent vessel occlusion, without simultaneous endosaccular coiling of the aneurysm, is the primary intent of the procedure
* Any absolute contraindication to endovascular treatment, angiography, or anaesthesia such as severe allergies to contrast or medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-11-13; Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Raymond, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (15):
- United States (8):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Stony Brook University Medical Center (SUNY), Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Virginia Health System, Charlottesville, Virginia
  - West Virginia University Hospital, Morgantown, West Virginia
- Canada (7):
  - Foothills Medical Center, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton General Hospital, Hamilton, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec

REFERENCES:
- [Background] White PM, Lewis SC, Gholkar A, Sellar RJ, Nahser H, Cognard C, Forrester L, Wardlaw JM; HELPS trial collaborators. Hydrogel-coated coils versus bare platinum coils for the endovascular treatment of intracranial aneurysms (HELPS): a randomised controlled trial. Lancet. 2011 May 14;377(9778):1655-62. doi: 10.1016/S0140-6736(11)60408-X. PMID 21571149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: November 2013 to june 2017, from 12 centres in Canada and U.S.A.
Period: Overall Study
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Started | 104 | 106
Completed | 99 | 95
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 3 | 4
Not completed — Death | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils | Total
Number analyzed (Participants) | 104 | 106 | 210
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10) | 57 (11) | 57 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 81 | 163
  Male | 22 | 25 | 47
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Major Recurrence of Lesion or Presence of Residual Aneurysm
Description: Major radiographic recurrence of the lesion or the presence of a 'residual aneurysm' as judged by core lab
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Number analyzed (Participants) | 104 | 106
Participants | 26 | 20

2. Primary Outcome: Hemorrhage During the Follow-up Period
Description: Post-treatment hemorrhage experienced during follow-up period.
Time Frame: Within 1 year following coiling
Measure: Count of Participants; unit: Participants
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Number analyzed (Participants) | 104 | 106
Participants | 0 | 1

3. Primary Outcome: Retreatment of the Same Lesion by Endovascular or Surgical Means
Description: Retreatment of the same lesion by endovascular or surgical means during the follow-up period
Time Frame: Within 1 year following coiling
Measure: Count of Participants; unit: Participants
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Number analyzed (Participants) | 104 | 106
Participants | 4 | 4

4. Primary Outcome: Initial Treatment Failure
Description: Inability to treat aneurysm, either because access to aneurysm is difficult or technical issues.
Time Frame: Within 1 year following coiling
Measure: Count of Participants; unit: Participants
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Number analyzed (Participants) | 104 | 106
Participants | 4 | 6

5. Primary Outcome: Related Morbidity
Description: Morbidity that precludes follow up
Time Frame: Within 1 year following coiling
Measure: Count of Participants; unit: Participants
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Number analyzed (Participants) | 104 | 106
Participants | 1 | 0

6. Secondary Outcome: Packing Density
Description: Packing density with the number of coils implanted
Time Frame: within the first 3 days after coiling
Measure: Mean (Standard Deviation); unit: percentage of packing density
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Number analyzed (Participants) | 100 | 99
percentage of packing density | 37.0 (22.2) | 26.9 (13.0)

7. Secondary Outcome: Procedural Serious Adverse Events (SAEs)
Description: Procedural-related serious adverse events
Time Frame: Within 6 months following coiling
Measure: Count of Participants; unit: Participants
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Number analyzed (Participants) | 104 | 106
Participants | 11 | 15

8. Secondary Outcome: Modified Rankin Score (mRS) Greater Than 2
Description: Modified Rankin Score (mRS) that is greater than 2 at 1 year follow-up (or at last follow-up, if applicable). Minimum = 0 (no symptoms), maximum = 6 (Deceased).
Time Frame: at 1 year follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Number analyzed (Participants) | 104 | 106
Participants | 3 | 7

9. Primary Outcome: Related Mortality
Description: Mortality that precludes follow up
Time Frame: Within 1 year following coiling
Measure: Count of Participants; unit: Participants
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
Number analyzed (Participants) | 104 | 106
Participants | 2 | 5

ADVERSE EVENTS:
Time Frame: Adverse Events are reported for a time period of within 1 year post aneurysm treatment.
Arm/Group | 15-caliber Platinum Coils | 10-caliber Coils
All-Cause Mortality (participants affected / at risk) | 2/104 | 7/106
Serious Adverse Events (participants affected / at risk) | 7/104 | 18/106
Other Adverse Events (participants affected / at risk) | 8/104 | 20/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 15-caliber Platinum Coils (N=104) | 10-caliber Coils (N=106)
Aneurysm rupture during procedure causing Mortality (Surgical and medical procedures) | 1 | 2
Stroke, periprocedure causing mortality (Vascular disorders) | 0 | 2
Stroke, related to SAH at presentation causing mortality (Vascular disorders) | 0 | 1
Subarachnoid hemorrhage during follow-up causing mortality (Vascular disorders) | 1 | 0
Event unrelated to aneurysm or its treatment causing mortality (General disorders) | 0 | 2
Aneurysm rupture during procedure causing morbidity (Surgical and medical procedures) | 3 | 4
Stroke, causing morbidity (Vascular disorders) | 2 | 6
SAH during follow-up, causing morbidity (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 15-caliber Platinum Coils (N=104) | 10-caliber Coils (N=106)
Hemorrhage (aneurysm rupture during procedure) (Vascular disorders) | 4 | 6
Stroke (Vascular disorders) | 2 | 11
Subarachnoid Hemorrhage during follow-up (Vascular disorders) | 1 | 1
Transient ischemic attack (TIA) (Vascular disorders) | 1 | 2

LIMITATIONS AND CAVEATS:
Trial was stopped before target number of patients were recruited due to funding being interrupted.

Premature interruption of the trial does not allow a conclusion regarding the primary hypothesis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than 12 months after the conclusion of the study at all sites.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT01943591/Prot_SAP_000.pdf